CLINICAL TRIAL: NCT04307160
Title: Effect of Age at Time of Surgery on the Surgical Outcome After Bilateral Lateral Rectus Muscle Recession in Intermittent Exotropia
Brief Title: Relationship of Age at Surgery to Surgical Outcome After Surgery for Intermittent Exotropia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Professor of Ophthalmology, Cairo University
Other Study IDs: D-31-2019
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients ≤ 5 years of age
  Interventions: Procedure: Bilateral lateral rectus recession
- Group II: Patients ≥ 7 years of age
  Interventions: Procedure: Bilateral lateral rectus recession

INTERVENTIONS:
Procedure: Bilateral lateral rectus recession — All patients will undergo bilateral lateral rectus recession according to standard tables. In the younger age group, the amount of lateral rectus recession will be reduced by 0.5 mm. in those with inferior oblique overaction, inferior oblique recession will be performed

SUMMARY:
It is prospective cohort study to compare ( the surgical outcome) the motor and sensory outcome of early surgery (≤5 years of age) and late surgery ( ≥ 7 years of age) for intermittent exotropia.

DETAILED DESCRIPTION:
Sample Size:

One hundred and twenty four patients with intermittent exotropia will be included in this study in form of two groups based on the age at the first surgery; each group including 62 patients

* Group I patients ≤ 5 years of age
* Group II patients ≥ 7 years of age

Sample size calculation:

We are planning a study of independent cases and controls with 1 control(s) per case. Prior data indicate that the success rate among adults is 0.75. If the success rate for the young age group is 0.5, we will need to study 58 adult subjects and 58 young subjects to be able to reject the null hypothesis that the success rates for young and adult subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. We will use an uncorrected chi-squared statistic to evaluate this null hypothesis. Assuming a dropout rate of 5 %, a total of 62 patients will be recruited in each group.

Inclusion criteria:

All patients with intermittent exotropia in whom surgery is indicated

Exclusion criteria:

Patients with prior eye muscle surgery, restrictive or paralytic strabismus will be excluded. In addition, patients with craniofacial anomalies or neurological problems will be excluded from the study.

Methodology (in details):

A detailed history will be obtained including presence of asthenopia, monocular closure, disfigurement or diplopia. The previous use of glasses for optical correction, use of minus lenses, or prior part time occlusion will be documented.

A detailed ophthalmological examination; including corrected and uncorrected visual acuity whenever feasible, cycloplegic refraction, anterior segment examination and dilated fundus examination for any abnormalities.

Motor Evaluation:

Ductions and versions will be done to assess the ocular motility in all diagnositic positions of gaze.

The angle of misalignment will be measured by the prism and alternate cover tests for both distance and near. The angle will be measured without and with glasses. The angles of misalignment will also be measured in side gazes and in straight up and down gaze whenever possible. In patients with near distance disparity, the angle of deviation will be measured again after patching one eye for 30 minutes, as well as after putting +3 D lenses in front of each eye.

The control of exotropia will be assessed using both the newcastle control score and the new intermittent exotropia control scale designed by Mohney and Holmes.

Sensory Evaluation:

TNO stereo test, titmus fly test and worth 4 dot test for far will be done whenever possible.

Surgery:

All patients will undergo bilateral lateral rectus recession according to standard tables. In the younger age group, the amount of lateral rectus recession will be reduced by 0.5 mm. in those with inferior oblique overaction, inferior oblique recession will be performed.

Follow up and Evaluation:

Postoperatively, patients will be examined in the same preoperative manner after one week then after 6 weeks, 3 month and 6 months to assess the horizontal alignment and do sensory evaluation whenever possible.

Statistical analysis:

Data management and analysis will be performed using Statistical Package for Social Sciences (SPSS) version (21). Median and range for non-parametric measures and ordinal (scores) data. Numerical data will be presented as means ± standard deviations (SD). Categorical data will be presented as number and percentages %. Pairwise comparisons between the two groups for normally distributed variables will be done using the Student's t-test; the Mann-Whitney test, a nonparametric test equivalent to the t-test, will be used in non-normally distributed variables. The pre and postoperative data will be compared using repeated measures ANOVA, with Friedman's test as its non-parametric equivalent. The chi-square test or the Fisher's exact test will be used to compare between the groups with respect to categorical data. All p-values will be two-sided. P-values < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

All patients with intermittent exotropia in whom surgery is indicated

Exclusion Criteria:

Patients with prior eye muscle surgery, restrictive or paralytic strabismus will be excluded. In addition, patients with craniofacial anomalies or neurological problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One hundred and twenty four patients with intermittent exotropia will be included in this study in form of two groups based on the age at the first surgery; each group including 62 patients
  * Group I patients ≤ 5 years of age
  * Group II patients ≥ 7 years of age Patients will be recruited from Kasr El Ainy and Cairo University Children Hospitals
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Motor success rate | Six months
  Success rate defined as deviation between exotropia/phoria of 8 PD to esotropia/phoria of 4 PD

SECONDARY OUTCOMES:
Change in stereoacuity | Six months
  Average log improvement of stereoacuity using TNO test at 6 months
New misalignment | Six months
  Number of patients who developed underaction, or overaction of horizontal or oblique muscles
Pattern deviation | Six months
  Number of patient who develop new A or V pattern after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Elshiaty, MD, Study Director — Head of Ophthalmology Department, Cairo University

REFERENCES:
- [Background] Buck D, Powell CJ, Sloper JJ, Taylor R, Tiffin P, Clarke MP; Improving Outcomes in Intermittent Exotropia (IOXT) Study group. Surgical intervention in childhood intermittent exotropia: current practice and clinical outcomes from an observational cohort study. Br J Ophthalmol. 2012 Oct;96(10):1291-5. doi: 10.1136/bjophthalmol-2012-301981. Epub 2012 Aug 11. PMID 22887975
- [Result] Richard JM, Parks MM. Intermittent exotropia. Surgical results in different age groups. Ophthalmology. 1983 Oct;90(10):1172-7. PMID 6657192
- [Result] Pratt-Johnson JA, Barlow JM, Tillson G. Early surgery in intermittent exotropia. Am J Ophthalmol. 1977 Nov;84(5):689-94. doi: 10.1016/0002-9394(77)90385-3. No abstract available. PMID 930997
- [Result] Haggerty H, Richardson S, Hrisos S, Strong NP, Clarke MP. The Newcastle Control Score: a new method of grading the severity of intermittent distance exotropia. Br J Ophthalmol. 2004 Feb;88(2):233-5. doi: 10.1136/bjo.2003.027615. PMID 14736781
- [Result] Abroms AD, Mohney BG, Rush DP, Parks MM, Tong PY. Timely surgery in intermittent and constant exotropia for superior sensory outcome. Am J Ophthalmol. 2001 Jan;131(1):111-6. doi: 10.1016/s0002-9394(00)00623-1. PMID 11162985
- [Result] Choi J, Kim SJ, Yu YS. Initial postoperative deviation as a predictor of long-term outcome after surgery for intermittent exotropia. J AAPOS. 2011 Jun;15(3):224-9. doi: 10.1016/j.jaapos.2010.12.019. Epub 2011 Jun 12. PMID 21665502
- See also: Changing patterns of strabismus: a decade of experience in Hong Kong — http://www.ncbi.nlm.nih.gov/pubmed/12140202
- See also: Binocular Vision and Ocular Motility THEORY AND MANAGEMENT OF STRABISMUS — http://www.aao.org/Assets/0c711d7f-503f-4cd9-b4ac-92d6ec31a718/636343503854270000/strabismus-binocular-vision-and-ocular-motility-vnoorden-pdf?inline=1